CLINICAL TRIAL: NCT01136135
Title: Cardiac MRI for the Detection of Cellular Rejection in Patients With Heart Transplantation
Brief Title: Cardiac Magnetic Resonance Imaging (CMRI) for Detection of Cardiac Transplant Rejection
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P081113; 2009-A00985-52 (Registry Identifier: ID RCB)
Record Dates: First submitted 2010-02-26; First posted 2010-06-03 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Heart Transplant Rejection
Keywords: Heart transplant rejection; cardiac MRI; diagnosis
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CARDIAC MRI
  Interventions: Other: CARDIAC MRI

INTERVENTIONS:
Other: CARDIAC MRI — To find a non-invasive alternative (with using cardiac MRI) to invasive endomyocardial biopsies for serial detection and follow-up of cellular rejection in heart transplant in childhood.

SUMMARY:
To find a non-invasive alternative (with using cardiac MRI) to invasive endomyocardial biopsies for serial detection (EMB) and follow-up of cellular rejection in heart transplant in childhood.

DETAILED DESCRIPTION:
Objectives To find a non-invasive alternative (with using cardiac MRI) to invasive endomyocardial biopsies for serial detection and follow-up of cellular rejection in heart transplant in childhood.

Background Detection of cardiac rejection is a major problem in cardiac transplantation. Invasive screenings at predefined time intervals for cellular rejection with using endomyocardial biopsies are standard procedures. However, cardiac biopsies are distressing and risky and are also costly. Moreover, as the histological expression of allograft rejection is patchy, endomyocardial biopsies may lead to sampling error. Thus, as the sensitivity is low and variable (range for 40 to 95%), indication of biopsy is still of debate.

Materials and methods All patients who undergone cardiac transplant are potentially eligible. They will be prospectively included in the study. They will have both examinations, their routine endomyocardial biopsies and cardiac MRI. Histological diagnosis of cellular rejection is given by the BILLINGHAM classification which is used in daily practice. Diagnosis of rejection of cardiac MRI is defined by the association of hyperintensity on T2-weighted sequence, and on gadolinium-enhanced sequences including SSFP (study state free precession) and myocardial delayed enhancement. Both MRI parameters attest of the presence of myocardial oedema related to acute rejection. Myocardial oedema is also associated with segmental abnormalities of myocardial contraction which is assessed by both CMR-tagged sequence.

Written informed consent will be required from the patients. Institutional review board approval will also be required.

Expected results and clinical implications We expect to demonstrate that CMRI is effective for detection of cellular rejection with a high sensitivity (expected sensitivity>95%) as compared to cardiac biopsy. In that condition, cardiac MRI could replace the invasive biopsy for serial detection and follow-up of rejection in heart transplant.

ELIGIBILITY:
Inclusion Criteria:

* all patients who had undergone cardiac transplants are eligible

Exclusion Criteria:

* no consent
* allergy to contrast agent (Gadolinium)
* severe renal failure (clearance < 30ml/min/1.73m²)
* claustrophobia
* severe arrhythmias
* absence of medical care insurance
* pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had undergone cardiac transplants
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2010-02; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The sensitivity and specificity of cardiac MRI for detecting heart transplant rejection will be calculated. The expected sensitivity and specificity are > 95%. | 24 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: Ou Phalla, MCU PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Necker, Paris, France